CLINICAL TRIAL: NCT03506295
Title: CrYobiopsy With Radial UltraSound Guidance (CYRUS)...
Brief Title: CrYobiopsy With Radial UltraSound Guidance
Acronym: CYRUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Fabien Maldonado, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 180058
Record Dates: First submitted 2018-03-07; First posted 2018-04-24 (Actual); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-10

CONDITIONS: Pulmonary Disease
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Primary bronchoscopist will perform localization of biopsy spot, after biopsy is determined to be in the control or intervention group. He/she will then perform the cryobiopsy per protocol. A bedside assistant will assist in managing the endobronchial blocker at all times. Secondary bronchoscopist will be stationed outside the operating room during initial part of the procedure. He will be prompted to enter the room by research coordinator to take control of the bronchoscope and assess post cryobiopsy bleeding. He will hence be blinded to the use or non-use of radial probe ultrasound. Research coordinator will be present at all times and will coordinate the switching process between proceduralists. Reference image of the radial USG determining the biopsy location on fluoroscopy monitor will be erased before secondary bronchoscopist enters the room. Patient will be blinded as he/she will be sedated. Four biopsies will be planned per procedure, two each from control & intervention arm.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control (Other): Standard of Care - Transbronchial cryobiopsies are obtained as a standard of care under fluoroscopy guidance
  Interventions: Device: Flouroscopy
- Intervention (Experimental): In the intervention arm , radial ultrasound probe will be used in addition to standard of care described above to confirm adequate position of the cryoprobe before transbronchial cryobiopsy is obtained.
  Interventions: Device: Radial Endobronchial Ultrasound Probe; Device: Flouroscopy

INTERVENTIONS:
Device: Radial Endobronchial Ultrasound Probe — The radial EBUS procedure is performed by inserting a miniature ultrasound probe (radial EBUS probe) through the working channel of a flexible bronchoscope or catheter (guide sheath). Real-time imaging of the surrounding tissue enables the clinician to determine the lesion's exact location and size.
  Arms: Intervention
Device: Flouroscopy — Real-time fluoroscopy will be used in all cases to guide the radial probe ultrasound and/or cryobiopsy probe placement.

SUMMARY:
Transbronchial cryobiopsy carries a higher chance of establishing pathological diagnosis in diffuse parenchymal lung disease (DPLD) than traditional transbronchial forceps guided biopsy. It is a novel technique capable of obtaining large, high-quality samples of lung tissue in a minimally invasive manner. This procedure may decrease the need for surgical lung biopsy in 75% of cases. However, there is an increased risk of pneumothorax and airway bleeding compared to traditional transbronchial forceps guided biopsy.

Several strategies are used by practitioners of this technique to mitigate the risks of significant bleeding and pneumothorax. These include prophylactic placement of an endobronchial blocker, the use of fluoroscopy guidance, instillation of cold saline to promote vasoconstriction, and establishment of a secure airway with endotracheal tube placement or rigid bronchoscopy

. Vanderbilt University Medical Center is one of the most active centers in terms of cryobiopsies performed as part of the diagnostic workup of DPLD. Currently all transbronchial cryobiopsies here are performed under fluoroscopic guidance, with endotracheal tube intubation and endobronchial blocker placement. Despite these precautions, post biopsy bleeding complications occur and can substantially lengthen the duration of the procedure and occasionally expose patients to procedural complications.

Radial ultrasound has been well utilized to define anatomy of peripheral lung and localization of peripheral pulmonary nodules. We postulate that using radial ultrasound to identify peribronchial lung parenchyma with low vascularity will mitigate the risk of hemorrhage during peripheral lung cryobiopsy in patients with DPLD and hence improve patient safety.

DETAILED DESCRIPTION:
Diffuse parenchymal lung diseases comprise a group of noninfectious, non-neoplastic lung diseases, each characterized by varying degrees of inflammation or fibrosis of the parenchyma of both lungs. The differentiation of these disorders may require biopsy material, particularly in patients with atypical clinical or radiological presentations. Cryobiopsies offer specialists the advantage of being able to collect much larger specimens than can be collected with forceps biopsy, while preserving the underlying lung architecture (no crush artifact). The biggest disadvantage of cryobiopsy is a higher risk of procedural bleeding and, to a lesser extent, pneumothorax than conventional transbronchial lung biopsies.

Existing cryobiopsy literature is significantly limited by lack of procedure standardization, variable diagnostic endpoints and non-uniform grading of complications. Surgical lung biopsy, currently the gold standard for histological diagnosis of DPLD, is associated with significant morbidity and mortality. The rate of in-hospital mortality following SLB for DPLD was recently found to be 1.7% in a large dataset, with a complication rate of 30% (including post-operative pneumothorax, pneumonia, respiratory failure). Mortality was slightly lower at 1.5% for elective operations but markedly higher at 16% for operations labeled "non-elective," presumably performed in the setting of acute disease exacerbations. Clearly, less invasive strategies, such as cryobiopsy, are urgently needed.

Recent studies demonstrate that there might be a trend toward more bleeding complications with transbronchial cryobiopsies. The increased risk of bleeding is due to the larger biopsies thus obtained, and the necessity to retrieve bronchoscope and cryoprobe en-bloc as biopsies are too large to be pulled through he working channel of the bronchoscope, preventing the proceduralist from keeping he bronchoscope wedged in the biopsied segment allowing bleeding tamponade. Accordingly, most proceduralists perform cryobiopsy with prophylactic placement of bronchial blocker positioned proximal to the selected lobe to occlude the segmental airway after biopsy. While this technique has essentially eliminated the risk of life-threatening bleeding after cryobiopsies, significant bleeding complications persist and can occasionally substantially lengthen the duration of the procedure, leading to premature termination and potentially quantitatively inadequate biopsy acquisition.

Conceptually it seems that the ability to select a less vascular area for a somewhat larger cryobiopsy may result in decreased risk of hemorrhage and/or reduction in bleeding severity. Average peripheral cryobiopsy size varies significantly and may be dependent on freezing time and cryoprobe size. Increase in resource utilization due to the use of radial ultrasound could be offset by a decrease in complication rate, decreased procedural time and potentially decreased endobronchial blocker need. This use of radial probe ultrasound use has not been widely reported in literature except for a recent single center retrospective review of 10 patients undergoing transbronchial cryobiopsies for ILD(Berim, 2017). Six of these patients underwent vascular localization with radial probe endobronchial localization with trends towards less bleeding.

The purported benefit of radial ultrasound-guided transbronchial cryobiopsy is the avoidance of excessive bleeding, which has been associated with this procedure. With the systematic use of a prophylactic bronchial blocker, an ideal endpoint for this pilot study would be the time spent obtaining each biopsy. We propose to study in a prospective, double-blind, randomized controlled fashion, the efficacy of radial endobronchial ultrasound (in combination with fluoroscopy) guided transbronchial cryobiopsy as compared to conventional fluoroscopy guided cryobiopsy in reducing time needed to achieve hemostasis (primary endpoint) and need for additional modalities to control bleeding and size of biopsies obtained (secondary endpoints).

ELIGIBILITY:
Inclusion Criteria:

1. Referral to interventional pulmonary services for diagnostic transbronchial cryobiopsy for diffuse parenchymal lung disease.
2. Transbronchial cryobiopsy is determined to be appropriately indicated as determined by consulting interventional pulmonologist.
3. Age > 18 years

Exclusion Criteria:

1. Inability to provide informed consent
2. Study subject has any condition that interferes with safe completion of the study including:

   1. Coagulopathy, with criteria left at the discretion of the operator
   2. Respiratory insufficiency with DLCO < 30% or baseline requirements of oxygen >2 liters
   3. Hemodynamic instability with systolic blood pressure <90 mmHg or heart rate > 120 beats/min, unless deemed to be stable with these values by the attending physicians
3. Patients representing vulnerable populations (prisoners, pregnant women, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Maldonado, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Each patient underwent TBC, and 4 samples of cryobiopsies were obtained per patient. 2 biopsies were obtained with Standard of Care procedures and 2 biopsies used the radial ultrasound probe will be used in addition to standard of care.
  All participants received both interventions.
Units Other Than Participants: cryobiopsies
Groups:
- All Participants: Each participant received 4 Transbronchial cryobiopsies during a single procedure:
  2 cryobiopsies are obtained as a standard of care under fluoroscopy guidance.
  The other 2 biopsies are obtained using a radial probe ultrasound under fluoroscopy guidance.
  All participants received both inventions during the same procedure.
  Fluoroscopy: Real-time fluoroscopy will be used in all cases to guide the radial probe ultrasound and/or cryobiopsy probe placement.
  fluoroscopy: Real-time fluoroscopy will be used in all cases to guide the radial probe ultrasound and/or cryobiopsy probe placement.
Period: Overall Study
Arm/Group | All Participants
Started | 10; 40 cryobiopsies
Completed | 10; 40 cryobiopsies
Not Completed | 0; 0 cryobiopsies

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants scheduled for cryobiopsy as part of their for routine clinical care had 4 biopsies: 2 with Transbronchial cryobiopsies as a standard of care and 2 with radial probe ultrasound. All participants received both interventions.
  Standard of Care - Transbronchial cryobiopsies are obtained as a standard of care under fluoroscopy guidance
  Fluoroscopy: Real-time fluoroscopy will be used in all cases to guide the radial probe ultrasound and/or cryobiopsy probe placement.
Arm/Group | All Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (9.789450104)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Time to Achieve Hemostasis After Obtaining Cryobiopsy
Description: This is defined as time from when the bronchoscope and cryoprobe are removed en bloc after obtaining the cryobiopsy to the time when it is determined to be safe to proceed to next cryobiopsy("Ready for next biopsy").
Time Frame: From time of randomization up to 120 minutes.
Population: All participants received both interventions during the same procedure.
Measure: Mean (Full Range); unit: seconds
Units Other Than Participants: biopsies
Groups:
- Control: Standard of Care - Transbronchial cryobiopsies are obtained as a standard of care under Fluoroscopy guidance
  fluoroscopy: Real-time Fluoroscopy will be used in all cases to guide the radial probe ultrasound and/or cryobiopsy probe placement.
- Intervention: In the intervention arm , radial ultrasound probe will be used in addition to standard of care described above to confirm adequate position of the cryoprobe before transbronchial cryobiopsy is obtained.
  Radial Endobronchial Ultrasound Probe: The radial EBUS procedure is performed by inserting a miniature ultrasound probe (radial EBUS probe) through the working channel of a flexible bronchoscope or catheter (guide sheath). Real-time imaging of the surrounding tissue enables the clinician to determine the lesion's exact location and size.
  Fluoroscopy: Real-time fluoroscopy will be used in all cases to guide the radial probe ultrasound and/or cryobiopsy probe placement.
Arm/Group | Control | Intervention
Number analyzed (Participants) | 10 | 10
Number analyzed (biopsies) | 20 | 20
seconds | 146.55 [7 to 614] | 132.25 [23 to 920]
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Other; p = 0.7878, Regression, Logistic; Odds Ratio (OR) = 0.496, 95% CI 2-sided [0.168 to 1.469]

2. Secondary Outcome: Grade of Bleeding
Description: 0)No or only scant bleeding, stops spontaneously
  1. Mild, stops with suction or iced saline or scope tamponade
  2. Modest, stops with balloon blockade < 3 min
  3. Moderate,requires bleeding side down in addition to balloon
  4. Severe, requires prolonged blockade (> 3 min)
  5. Very severe,soils opposite lung, hypoxemia, increase level of care, additional procedures All participants received both interventions during the same procedure.
Time Frame: From time of randomization up to 120 minutes.
Population: All participants received both interventions during the same procedure.
Measure: Count of Units; unit: cryobiopsies
Units Other Than Participants: cryobiopsies
Arm/Group | Control | Intervention
Number analyzed (Participants) | 10 | 10
Number analyzed (cryobiopsies) | 20 | 20
cryobiopsies
  0)No or only scant bleeding, stops spontaneously | 9 | 12
  1)Mild, stops with suction or iced saline or scope | 8 | 7
  2) Modest, stops with balloon blockade < 3 min | 2 | 1
  3)Moderate,requires bleeding side down in addition | 0 | 0
  4) Severe, requires prolonged blockade (> 3 min) | 1 | 0
  5)Very severe,soils opposite lung, hypoxemia, incr | 0 | 0

3. Secondary Outcome: Number of Biopsies That Required Additional Interventions to Manage Bleeding
Description: Cold saline, patient positioning, rigid bronchoscopy, embolization, ICU admission etc. are techniques to control bleeding after cryobiopsy. Use of these techniques will be recorded.
Time Frame: From time of randomization up to 120 minutes.
Population: All participants received both interventions during the same procedure.
Measure: Number; unit: biopsies
Units Other Than Participants: cryobiopsies
Arm/Group | Control | Intervention
Number analyzed (Participants) | 10 | 10
Number analyzed (cryobiopsies) | 20 | 20
biopsies | 6 | 5

4. Secondary Outcome: Biopsy Specimen Quality
Description: Each biopsy obtained will be assessed by pathologist for quality of sample obtained and injury patterns identified
Time Frame: From time of randomization until acquisition of results from pathology, assessed up to 12 months.
Population: this analysis was removed from the protocol and data were not collected
Units Other Than Participants: crypbiopsies
Arm/Group | Control | Intervention
Number analyzed (Participants) | 0 | 0
Number analyzed (crypbiopsies) | 0 | 0

5. Secondary Outcome: Biopsy Size
Description: Each biopsy obtained will be assessed by pathologist for size of sample obtained.
Time Frame: From time of randomization until acquisition of results from pathology, assessed up to 12 months.
Population: this analysis was removed from the protocol and data were not collected
Units Other Than Participants: crypbiopsies
Arm/Group | Control | Intervention
Number analyzed (Participants) | 0 | 0
Number analyzed (crypbiopsies) | 0 | 0

ADVERSE EVENTS:
Time Frame: The perioperative period until discharge. (24 hours)
Description: Definition of adverse event and/or serious adverse event, used to collect adverse event information does not differ from the clinicaltrials.gov.
Groups:
- All Participants: All participants received both interventions during the same procedure:
  2 biopsies via Standard of Care - Transbronchial cryobiopsies are obtained as a standard of care under fluoroscopy guidance
  2 biopsies via Radial Probe Ultasound - Transbronchial cryobiopsies are obtained with a Radial Probe Ultasound under fluoroscopy guidance
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
1. Considering the difference in thickness and flexibility of cryoprobe as compared to REBUS probe, thei positioning may not always truly coincide.
2. Operator dependent observer's bias while obtaining hemostasis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/95/NCT03506295/Prot_SAP_000.pdf